CLINICAL TRIAL: NCT01528865
Title: A Phase I/II Study of Safety and Efficacy of Lamivudine (EPIVIR®) and Tenofovir Disoproxil Fumarate (VIREAD®) Used to Lower the Plasma Level of Viral RNA of HERV-K(HML2) in Patients With Lymphoma
Brief Title: Safety & Efficacy of Lamivudine & Tenofovir to Lower Plasma Level of Viral RNA in Lymphoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding was removed.
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UMCC 2010 097; HUM 33361 (Other: University of Michigan IRBMED)
Record Dates: First submitted 2012-01-12; First posted 2012-02-08 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Lymphoma
Keywords: virus; K(HML2)[HERV-K(HML2)]; Lymphoma; Human endogenous retrovirus-K(HLM2)[HERV-K(HML2)]
MeSH Terms: conditions — Lymphoma; Virus Diseases | interventions — Lamivudine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Drugs (Experimental): The medications to be used in this study are Lamivudine (EPIVIR®) and Tenofovir disoproxil fumarate (VIREAD®), medications already used in people with certain other types of viruses [but not HERV-K(HML2)] in their body. Treatment will last 16 weeks. This is an experiment combining these two drugs and has been issue an Investigational New Drug (IND) Exemption by the FDA.
  Interventions: Drug: Lamivudine; Drug: Tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Lamivudine — Creatinine Clearance (mL/min): ≥50, Recommended Dosage of Epivir: 150 mg twice daily or 300 mg once daily.
  Creatinine Clearance (mL/min): 30-49, Recommended Dosage of Epivir: 150 mg once daily.
  Subjects will be taking drug for 16 weeks.
  Other Names: Epivir
Drug: Tenofovir disoproxil fumarate — 300 mg once a day p.o. for 16 weeks.
  Other Names: Viread

SUMMARY:
Therapy for non-Hodgkin lymphoma (NHL) is in evolution as new molecular pathways and targeted therapies are identified. Although most NHLs respond to currently available therapies, the majority of patients relapse and many never have a complete response to therapy. In the investigators attempts to further understand the pathogenesis of NHLs, the investigators have identified and characterized expression of human endogenous retroviruses (HERVs) at the DNA, RNA and protein levels in association with the presence of NHLs (and other neoplastic diseases). The investigators preclinical evidence suggests a correlation with the level of HERV-K (a particular family of HERVs) expression and NHL disease activity, leading us to hypothesize that HERV-K expression may contribute to the development of the disease and/or to its recurrence. If this hypothesis is correct, then drugs that inhibit HERV-K expression may prevent recurrence of disease and/or may provide a novel therapeutic approach for NHLs.

To test this hypothesis, the investigators eventually intend to study the use of anti-retroviral therapies in patients with NHL. The investigators in vitro studies have demonstrated that HERV-K expression decreases in response to the currently FDA-approved and available, anti-HIV drugs, Lamivudine and tenofovir disoproxil fumarate (tenofovir). These medications are tolerated well in HIV patients, but it is unknown how the combination of Lamivudine and Tenofovir will be tolerated by patients with NHL. To further test the investigators hypotheses, the investigators propose the following Specific Aims of the current study: (1) To evaluate the tolerability, toxicity and safety of administering Lamivudine and Tenofovir in combination to patients with relapsed or refractory NHL; (2) To evaluate the effects of the combination of lamivudine and tenofovir on HERV-K plasma viral RNA load; and (3) To monitor the response rate of the NHL to treatment with the combination of lamivudine and tenofovir.

The investigators study will recruit adult patients with relapsed or refractory NHL whom the investigators have identified as having expression of HERV-K. Volunteer participants will be administered the combination of lamivudine and tenofovir and monitored for tolerability, toxicity, compliance, changes in viral RNA load and disease response.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of non-Hodgkin lymphoma (NHL)
* Must have HERV-K(HML2) viral load of ≥1x103 using a gag primer reverse transcriptase polymerase chain reaction (RT-PCR) assay.
* Must have bi-dimensionally measurable disease.
* Patients with lymphomas that are felt to be incurable with any therapy and for whom there are no standard treatments that would be anticipated to be necessary or beneficial within the next 5 months. These patients can have received any amount of prior chemotherapy to enter this trial.
* All previous therapies must have been discontinued at least 4 weeks prior to initiation of the administration of this study's drugs.
* HIV negative by standard blood testing.
* Have an expected life expectancy of at least 5 months.
* Have an Eastern Cooperative Oncology Group (ECOG) performance scale status of 0 - 2l) Must have a serum creatinine <2.0 and creatinine clearance >30 ml/min/m2. Other organ dysfunction is eligible at the discretion of the PI.
* Agree to use a reliable method of birth control prior to drug initiation and for the duration of their study participation.

Exclusion Criteria:

* a) Have received chemotherapy or radiotherapy within 4 weeks
* Have not recovered from the adverse effects or toxicities of lymphoma therapy most recently administered.
* Currently receiving any other investigational medication or therapy.
* Patients with a second malignancy that might interfere with interpretation of the results of this study.
* Patients with known allergic reaction to lamivudine or tenofovir disoproxil fumarate (DF).
* Patients on drugs that interfere with renal function or drugs that compete with tenofovir for active binding sites (i.e. intravenous cidofovir, acyclovir, ganciclovir, and valganciclovir).
* Uncontrolled concurrent illnesses, including, but not limited to, active/ongoing infection, symptomatic congestive heart failure, unstable angina pectoris.
* Women who are pregnant, become pregnant, or are breast-feeding.
* Standard blood tests that are positive for HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy (effect on human endogenous retrovirus-K(HML2)[HERV-K(HML2)] | 2 years
  Patients will have HERV-K(HML2) viral load measured at baseline and post-treatment (quantifiable HERV-K(HML2) viral load is an eligibility criterion, and post-treatment loads below the limit of quantitation will be assigned a random value uniformly distributed between 0 and the limit of quantitation).

SECONDARY OUTCOMES:
tumor regression | 2 years
  Linear models will be used to relate tumor regression to change in viral load of RNA levels.
Toxicity will be tabulated according to NCI NCI Common Terminology Criteria for Adverse Events (CTCAE) v4 grade and classification | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States